CLINICAL TRIAL: NCT03650244
Title: Nationwide Observation Study to Evaluate the Efficacy and Tolerance of the Adjustable Medical Device REMEEX® in the Treatment of Male Stress Urinary Incontinence
Acronym: Remeex
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2016/LW-01
Record Dates: First submitted 2017-06-30; First posted 2018-08-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients fitted with REMEEX
  Interventions: Device: REMEEX implantation

INTERVENTIONS:
Device: REMEEX implantation — Device implantation

SUMMARY:
We wish to set up a multicentric prospective observational study across France to collate data on the efficacy and tolerance of the Male REMEEX® device in patients with moderate stress urinary incontinence following radical prostatectomy. Patient satisfaction, improvement in quality of life, side effects and complications will also be studied, as will the ease of use of the device from the point of view of the surgeon. A long-term follow-up of 5 years will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been informed about the study
* The patient is at least 18 years old
* Patient suffering from moderate stress incontinence (pure or predominant) following radical prostatectomy surgery, for at least 12 months, unresolved after of pelvic floor reeducation
* Patient scheduled for REMEEX® implant

Exclusion Criteria:

* It proves impossible to give the patient clear information
* Patient refuses to participate
* Life expectancy of the patient estimated to be less than the 5 year follow-up
* Impossible to contact patient after hospitalization
* Radiotherapy of less than 6 month
* Patient unable to fill in questionnaire
* Incapably of performing pad test at 24 hours
* Recurrent symptomatic prostate cancer
* Mixed incontinence with urgency incontinence
* Bladder outlet obstruction: stenosis of the vesico-urethral anastomosis or untreated urethral stricture.
* Post void residual >100ml
* Other cancer under treatment or progressing
* Kidney injury, hepatocellular insufficiency
* Auto-immune disease
* Neurological-origin urinary incontinence (stroke, MS, Parkinson's)
* Incontinence arising from surgery other than prostatectomy
* recurrent gross hematuria
* Recurrent urinary infection
* Bladder stones

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 suffering from moderate stress incontinence (pure or predominant) following radical prostatectomy surgery for prostate cancer, for at least 12 months, unresolved after of pelvic floor reeducation, regardless of the surgical procedure used or of treatment with radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11-16 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficacy of REMEEX® on urinary incontinence post radical prostatectomy | 1 month
  PAD test < 2 g / 24 h
Evaluate efficacy of REMEEX® on urinary incontinence post radical prostatectomy | 6 months
  PAD test < 2 g / 24 h
Evaluate efficacy of REMEEX® on urinary incontinence post radical prostatectomy | 1 year
  PAD test < 2 g / 24 h
Evaluate efficacy of REMEEX® on urinary incontinence post radical prostatectomy | 2 years
  PAD test < 2 g / 24 h
Evaluate efficacy of REMEEX® on urinary incontinence post radical prostatectomy | 3 years
  PAD test < 2 g / 24 h
Evaluate efficacy of REMEEX® on urinary incontinence post radical prostatectomy | 4 years
  PAD test < 2 g / 24 h
Evaluate efficacy of REMEEX® on urinary incontinence post radical prostatectomy | 5 years
  PAD test < 2 g / 24 h

SECONDARY OUTCOMES:
Normal clinical examination | month 1
  Yes / No
Normal clinical examination | Month 6
  Yes / No
Normal clinical examination | Year 1
  Yes / No
Normal clinical examination | Year 2
  Yes / No
Normal clinical examination | Year 3
  Yes / No
Normal clinical examination | Year 4
  Yes / No
Normal clinical examination | Year 5
  Yes / No
urinary output | Month 1
  ml/s
urinary output | Month 6
  ml/s
urinary output | year 1
  ml/s
urinary output | year 2
  ml/s
urinary output | year 3
  ml/s
urinary output | year 4
  ml/s
urinary output | year 5
  ml/s
Volume of urine | month 1
  ml
Volume of urine | month 6
  ml
Volume of urine | year 1
  ml
Volume of urine | year 2
  ml
Volume of urine | year 3
  ml
Volume of urine | year 4
  ml
Volume of urine | year 5
  ml
Post-void residual urine volume | Month 1
  ml
Post-void residual urine volume | Month 6
  ml
Post-void residual urine volume | year 1
  ml
Post-void residual urine volume | year 2
  ml
Post-void residual urine volume | year 3
  ml
Post-void residual urine volume | year 4
  ml
Post-void residual urine volume | year 5
  ml
cystoscopy | Month 1
  Yes / No
cystoscopy | Month 6
  Yes / No
cystoscopy | year 1
  Yes / No
cystoscopy | year 2
  Yes / No
cystoscopy | year 3
  Yes / No
cystoscopy | year 4
  Yes / No
cystoscopy | year 5
  Yes / No
readjustment of the REMEEX medical device | Month 1
  Yes / No
readjustment of the REMEEX medical device | Month 6
  Yes / No
readjustment of the REMEEX medical device | Year 1
  Yes / No
readjustment of the REMEEX medical device | Year 2
  Yes / No
readjustment of the REMEEX medical device | Year 3
  Yes / No
readjustment of the REMEEX medical device | Year 4
  Yes / No
readjustment of the REMEEX medical device | Year 5
  Yes / No
General improvement of symptoms | 1 month
  Patient Global Impression of Improvement Questionnaire (PGI-I)
General improvement of symptoms | 6 months
  Patient Global Impression of Improvement Questionnaire (PGI-I)
General improvement of symptoms | 1 year
  Patient Global Impression of Improvement Questionnaire (PGI-I)
General improvement of symptoms | 2 years
  Patient Global Impression of Improvement Questionnaire (PGI-I)
General improvement of symptoms | 3 years
  Patient Global Impression of Improvement Questionnaire (PGI-I)
General improvement of symptoms | 4 years
  Patient Global Impression of Improvement Questionnaire (PGI-I)
General improvement of symptoms | 5 years
  Patient Global Impression of Improvement Questionnaire (PGI-I)
Improvement of urinary symptoms | 1 month
  Urinary Symptom Profile Questionnaire (USP)
Improvement of urinary symptoms | 6 months
  Urinary Symptom Profile Questionnaire (USP)
Improvement of urinary symptoms | 1 year
  Urinary Symptom Profile Questionnaire (USP)
Improvement of urinary symptoms | 2 years
  Urinary Symptom Profile Questionnaire (USP)
Improvement of urinary symptoms | 3 years
  Urinary Symptom Profile Questionnaire (USP)
Improvement of urinary symptoms | 4 years
  Urinary Symptom Profile Questionnaire (USP)
Improvement of urinary symptoms | 5 years
  Urinary Symptom Profile Questionnaire (USP)
Side effects or complications | 1 month
Side effects or complications | 6 months
Side effects or complications | 1 year
Side effects or complications | 2 years
Side effects or complications | 3 years
Side effects or complications | 4 years
Side effects or complications | 5 years
Reliability and ease of use of the device | 1 month
Reliability and ease of use of the device | 6 months
Reliability and ease of use of the device | 1 year
Reliability and ease of use of the device | 2 years
Reliability and ease of use of the device | 3 years
Reliability and ease of use of the device | 4 years
Reliability and ease of use of the device | 5 years
Patient incontinence-related quality of life | 1 month
  Incontinence Quality of Life Questionnaire (I-QOL)
Patient incontinence-related quality of life | 6 months
  Incontinence Quality of Life Questionnaire (I-QOL)
Patient incontinence-related quality of life | 1 year
  Incontinence Quality of Life Questionnaire (I-QOL)
Patient incontinence-related quality of life | 2 years
  Incontinence Quality of Life Questionnaire (I-QOL)
Patient incontinence-related quality of life | 3 years
  Incontinence Quality of Life Questionnaire (I-QOL)
Patient incontinence-related quality of life | 4 years
  Incontinence Quality of Life Questionnaire (I-QOL)
Patient incontinence-related quality of life | 5 years
  Incontinence Quality of Life Questionnaire (I-QOL)
Patient sexual-related quality of life | 1 month
  International Index of Erectile Function (IIEF-5) score
Patient sexual-related quality of life | 6 months
  International Index of Erectile Function (IIEF-5) score
Patient sexual-related quality of life | 1 year
  International Index of Erectile Function (IIEF-5) score
Patient sexual-related quality of life | 2 years
  International Index of Erectile Function (IIEF-5) score
Patient sexual-related quality of life | 3 years
  International Index of Erectile Function (IIEF-5) score
Patient sexual-related quality of life | 4 years
  International Index of Erectile Function (IIEF-5) score
Patient sexual-related quality of life | 5 years
  International Index of Erectile Function (IIEF-5) score
Satisfaction of use by the surgeon. | Day 0
  anological visual scale (between 0 and 10)

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU de Besançon, Besançon
  - APHP Hôpital Henry Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Limoges, Limoges
  - CHU Nancy, Nancy
  - CHU Nice, Nice
  - CHU Nimes, Nîmes
  - CHU Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No